CLINICAL TRIAL: NCT02653352
Title: School Randomised Trial on Prevention of Excessive Weight Gain by Discouraging Students From Drinking Sodas
Brief Title: Prevention of Excessive Weight Gain by Discouraging Students From Drinking Sodas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rio de Janeiro State University (Other)
Collaborators: National Research Council, Brazil (Other); Universidade Federal do Rio de Janeiro (Other)
Responsible Party: Principal Investigator, Rosely Sichieri, Professor, Rio de Janeiro State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 500404/2003-8
Record Dates: First submitted 2015-11-23; First posted 2016-01-12 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2015-11

CONDITIONS: Overweight; Children
Keywords: randomized controlled trials; soft drinks; hypercholesterolemia; serum cholesterol; blood glucose; overweight; carbonated beverages
MeSH Terms: conditions — Overweight; Hypercholesterolemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): The control group received two one-hour general sessions on health issues and printed general advices regarding healthy diets.
- Lifestyle modification (Experimental): Intervention was focused on the reduction in consumption of sugar-sweetened carbonated beverages by students. During seven months of one school year, a healthy lifestyle education programme was implemented using simple messages encouraging water consumption instead of sugar-sweetened carbonated beverages. Education was delivered via classroom activities; banners were hung promoting water consumption, and water bottles with the logo of the campaign were given to children and schoolteachers.
  Interventions: Behavioral: Lifestyle modification

INTERVENTIONS:
Behavioral: Lifestyle modification — The centre of the campaign was to encourage the exchange of sugar-sweetened beverages for water. Ten one-hour sessions of activities facilitated by four trained research assistants were assigned for each class. The activities required 20-30 min and teachers were encouraged to reiterate the message during their lesson. Classroom quizzes and games using water v. sugar-sweetened carbonated beverages as the theme, as well as song and drawing competitions, were promoted. In addition, a musician using a tambourine helped each class to collectively develop songs related to drinking water and reducing the consumption of sugar-sweetened carbonated beverages. This musical activity was conducted during three one-hour sessions.
  Arms: Lifestyle modification

SUMMARY:
The purpose of this study was to encourage students to reduce soft drinks intake, substituting it by water, in order to prevent and control overweight prevalence.

DETAILED DESCRIPTION:
During seven months of one school year, a healthy lifestyle education programme was implemented using simple messages encouraging water consumption instead of sugar sweetened carbonated beverages. The messages were previously tested for understanding in two small groups of children of the same age and socio-economic background as the study participants. Also, beliefs and behaviors of children in these focus groups were recorded in order to orient activities and the production of printed materials to be given to participants. Education was delivered via classroom activities; banners were hung promoting water consumption, and water bottles with the logo of the campaign were given to children and schoolteachers.

ELIGIBILITY:
Inclusion Criteria:

* 4th grade morning classes

Exclusion Criteria:

* Pregnancy
* Physical disabilities preventing anthropometric measurement

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1140 (Actual)
Dates: Start 2005-03; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Change in body mass index (kg/m²) | baseline, 8 months
  We have calculated changes in body mass index (BMI in follow-up minus BMI on baseline) and compared mean changes between control and intervention groups, in order to address differences in BMI gain among groups.

SECONDARY OUTCOMES:
Change in overweight prevalence as assessed by percentage of overweight participants | baseline, 8 months
  Prevalence of overweight was assessed in both groups (intervention and control) in baseline and at the end of follow-up, according to standard definition proposed by Cole et al., 2000. Then, we evaluated changes in prevalences among groups.
Change in obesity prevalence as assessed by percentage of obese participants | baseline, 8 months
  Prevalence of obesity was assessed in both groups (intervention and control) in baseline and at the end of follow-up, according to standard definition proposed by Cole et al., 2000. Then, we evaluated changes in prevalences among groups.
Change in blood cholesterol | baseline, 8 months
Change in blood glucose | baseline, 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Rosely Sichieri, PhD, Principal Investigator — State University of Rio de Janeiro

REFERENCES:
- [Background] Schulze MB, Manson JE, Ludwig DS, Colditz GA, Stampfer MJ, Willett WC, Hu FB. Sugar-sweetened beverages, weight gain, and incidence of type 2 diabetes in young and middle-aged women. JAMA. 2004 Aug 25;292(8):927-34. doi: 10.1001/jama.292.8.927. PMID 15328324
- [Background] Malik VS, Pan A, Willett WC, Hu FB. Sugar-sweetened beverages and weight gain in children and adults: a systematic review and meta-analysis. Am J Clin Nutr. 2013 Oct;98(4):1084-102. doi: 10.3945/ajcn.113.058362. Epub 2013 Aug 21. PMID 23966427
- [Result] Sichieri R, Paula Trotte A, de Souza RA, Veiga GV. School randomised trial on prevention of excessive weight gain by discouraging students from drinking sodas. Public Health Nutr. 2009 Feb;12(2):197-202. doi: 10.1017/S1368980008002644. Epub 2008 Jun 18. PMID 18559131
- [Result] Vargas IC, Sichieri R, Sandre-Pereira G, da Veiga GV. Evaluation of an obesity prevention program in adolescents of public schools. Rev Saude Publica. 2011 Feb;45(1):59-68. doi: 10.1590/s0034-89102011000100007. English, Portuguese. PMID 21181050